CLINICAL TRIAL: NCT01554592
Title: Polypharmacy in the Heart Failure Patient: Are All Prescribed Drug Classes Required? Statin Withdrawal Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Dr Ingrid Hopper, The Alfred
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP-02/12
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Statin withdrawal
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin withdrawal (Experimental): Participants will received a placebo for 12 weeks.
  Interventions: Drug: Withdrawal of statin therapy
- Stable statin therapy (Active Comparator): Participants need to have been receiving statin therapy for at least 3 months and be on a stable dose.
  Interventions: Drug: Statin therapy

INTERVENTIONS:
Drug: Withdrawal of statin therapy — Participants currently received statin therapy will have their statin stopped for 12 weeks.
  Arms: Statin withdrawal
Drug: Statin therapy — Participants will continue on stable statin therapy.
  Arms: Stable statin therapy

SUMMARY:
Heart failure (cardiomyopathy) is a chronic condition in which the heart fails to function as a pump to move blood around the body. This sets up a complex physiologic response to compensate, which include activation of many hormonal mechanisms which result in fluid accumulation.

In recent years, medications to block the hormonal response to heart failure are given as standard drugs, and these include ACE inhibitors and beta blockers. Mortality is reduced with these medications, as well as symptoms improved. Other medications are also used in heart failure, for which a clear-cut benefit has not been demonstrated. Statins, also called HMG CoA reductase inhibitors, are used to reduce cholesterol levels and can help to prevent heart failure by preventing heart attacks. They have been used in heart failure that is not caused by heart attacks in the belief that they had "pleiotropic" effects, meaning that they had beneficial effects in heart failure separate from the reduction in cholesterol.

However large trials in heart failure have demonstrated that statins do not increase survival compared with placebo. There is no evidence to recommend their routine use in established heart failure caused by either heart attacks or genetics.

The investigators propose that the use of statins in heart failure is unnecessary and could be stopped. The importance of finding evidence to cease unproven medications in heart failure cannot be understated. Patients with heart failure take an average of six prescription medications each day. Each medication has side effects and the interactions of all the drugs together are unknown. Statins are the commonest reason for side effects in patients with heart failure, causing muscle pains and gastrointestinal upset.

In this study, the investigators plan to withdraw statins from patients with stable heart failure in a closely monitored environment and watch for the effect of this on heart failure and on how they feel generally.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years
2. Documented heart failure of ischaemic, idiopathic or hypertensive cause
3. New York Heart Association (NYHA) class II, III or IV symptoms
4. LVEF < 0.40, or no more than 0.35 if NYHA class II and ischaemic aetiology.
5. Receiving ACE inhibitor or ARB (Angiotensin II Receptor Blockers), β-blocker and diuretic therapy at the optimal doses.
6. Has been receiving statin therapy for at least 3 months
7. Willing and able to provide informed consent

Exclusion Criteria:

1. Treatment with statins primarily for treatment of hypercholesterolaemia
2. Obstructive or restrictive cardiomyopathy
3. Uncorrected primary valvular disease
4. Active myocarditis
5. Decompensated heart failure or a need for inotropic therapy
6. Myocardial infarction within the past 6 months
7. Unstable angina or stroke within the past 3 months
8. PCI (Percutaneous coronary intervention), CABG (coronary artery bypass graft)or implantation of cardioverter-defibrillator or biventricular pacemaker within the past 3 months or a planned implantation of such a device
9. Previous or planned cardiac transplantation
10. Pericardial disease or systemic disease (eg amyloidosis)
11. Acute or chronic liver disease
12. Alanine and aspartate transminase concentrations more than 1.5 times the upper limit of normal
13. Chronic muscle disease or an unexplained creatinine kinase level of more than 2.5 times the upper limit of normal
14. Serum creatinine level greater than 221 micromol/L
15. Previous treatment with cyclosporine
16. Exercise capacity limited by factors other than cardiac dyspnoea
17. Hospitalisation within one month of randomisation
18. Pregnant or lactating women or women of childbearing potential who were not adequately protected against becoming pregnant
19. Any other concurrent condition that, in the opinion of the investigator, would prevent completion of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
NYHA (New York Heart Association) Heart Failure class | baseline and after 12 weeks of treatemnt

SECONDARY OUTCOMES:
6 minutes walk test | Baseline and after 12 weeks of treatment
Quality of life questionnaire | Baseline and after 12 weeks of treatment
Change in BNP (Brain natriuretic peptide) | Baseline and after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Alfred Hospital/Monash University
Locations (1):
- Clinical Pharmacology, Alfred Hospital, Melbourne, Victoria, Australia